CLINICAL TRIAL: NCT03336307
Title: Predictors of Gait Improvement in Patients With Parkinson's Disease After Rehabilitation
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mariano Serrao, Clinical Professor, University of Roma La Sapienza
Other Study IDs: s001
Record Dates: First submitted 2017-10-10; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease; Movement Disorders
Keywords: Parkinson disease; movement Disorders; gait disturbance; Parkinson; Parkinson gait; 3D motion analysis systems; motion analysis; Parkinson rehabilitation; rehabilitation gait improvement; gait improvement; SMART Capture; MATLAB software
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Mobility Limitation | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Parkinson's disease: All participants could walk independently without walking devices. All patients were taking oral administrations of levodopa (18 patients), dopamine agonists (5 patients), or both (13 patients) and were recorded in on phase. Medication was kept constant throughout the trial, and all interventions were performed at the same time of day for each patient during ON phase.
  Severity of parkinsonism was evaluated using the Unified Parkinson's Disease Rating Scale (UPDRS-II and III) and the Hoehn and Yahr staging system.
  All patients received a rehabilitation program planned according to the European Physiotherapy guideline for Parkinson's disease
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — all patients received a rehabilitation program planned according to the European Physiotherapy guideline for Parkinson's disease and focus on:
  * endurance, strength, flexibility and balance with functional practice for all H/Y stage
  * endurance also for H/Y stage 1,
  * motor learning principles and cue functional for H/Y stage 2-3
  * external cues and self-instruction strategies and attention H/Y for stage 2-3 The rehabilitative program comprised 60-minute sessions a day (3d/wk).

SUMMARY:
Patients with Parkinson's disease show a gait disturbance which is considered as one of the most disabling aspect of the disease that strongly impacts on patients' autonomy and quality of life. The mechanism underlying gait impairment is multi-factorial, reflects the global motor impairment of patients with PD and is mainly related to a neurotransmitter deficiency inducing bradykinesia, rigidity, abnormal trunk control and postural instability. For this reason, and considering the impact of social and economic costs, one of the main foci of intervention in patients with PD should be treating gait abnormalities. This need is further reinforced by the knowledge that gait outcomes are correlated with longevity, cognitive decline and adverse events.

Besides the shorten-step gait clinical description of the gait disorder in PD, in the last years, studies using modern 3D motion analysis systems have further detailed the gait pattern in PD disclosing abnormalities in cadence, stance duration, swing duration, double support duration, leg length, step length, velocity, hip, knee and ankle ROMs. Such abnormal gait parameters seem to correlate with the clinical outcomes of UPDRS score, H-Y stage and milliequivalents of levodopa taken. Importantly, gait parameters can either normalize or improve after several rehabilitative treatment strategies including physiotherapy, assistive equipment, sensory cueing, treadmill training, physical activity, home base exercises. However, none of the previous studies specifically investigated which biomechanical factor can be modified after rehabilitation and which clinical characteristic can predict the rehabilitation-induced gait improvement. This would be extremely important to typifying, grouping and selecting patients, optimizing the rehabilitative strategies and cost management.

The aims of the present study were to evaluate in a sample of patients with PD: i) which gait parameters can be modified after a short-term rehabilitation program; ii) which, if any, clinical variable can predict the improvement of the gait function after rehabilitation. At this aim we quantitatively evaluated the gait performance of PD patients by means of a 3-D motion analysis system.

DETAILED DESCRIPTION:
Fifty out of 67 patients with idiopathic PD assessed for eligibility were recruited at Rehabilitation Unit of Department of Medical and Surgical Sciences and Biotechnologies, University of Rome, Sapienza, and at Rehabilitation Unit of Policlinico Italia Centre, Rome, Italy. Patients were admitted for outpatient rehabilitation between May 2014 and April 2017. The inclusion criteria were a diagnosis of idiopathic PD according to UK bank criteria and Hoehn and Yahr stages 1 to 3. All patients were in a stable drug program and had adapted to their current medications for at least 2 weeks. Exclusion criteria were: cognitive deficits (defined as scores of <26 on the Mini-Mental State Examination [MMSE]), moderate or severe depression (defined as scores of >17 on the Beck Depression Inventory [BDI]), and orthopedic and other gait-influencing diseases such as arthrosis or total hip joint replacement.

All participants could walk independently without walking devices. All patients were taking oral administrations of levodopa (18 patients), dopamine agonists (5 patients), or both (13 patients) and were recorded in on phase.

Severity of parkinsonism was evaluated using the Unified Parkinson's Disease Rating Scale (UPDRS-II and III) and the Hoehn and Yahr staging system.

The study complied with the Helsinki Declaration and received local ethics committee approval. Prior to taking part in the study, all the participants gave a written consent after a fully explanation of the experimental procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD according to UK bank criteria
* Hoehn and Yahr stages 1 to 3.
* All patients were in a stable drug program and had adapted to their current medications for at least 2 weeks

Exclusion Criteria:

* Cognitive deficits (defined as scores of <26 on the Mini-Mental State Examination [MMSE]),
* moderate or severe depression (defined as scores of >17 on the Beck Depression Inventory [BDI]), -. orthopedic and other gait-influencing diseases such as arthrosis or total hip joint replacement.

Ages: 48 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty out of 67 patients with idiopathic PD assessed for eligibility were recruited at Rehabilitation Unit of Department of Medical and Surgical Sciences and Biotechnologies, University of Rome, Sapienza, and at Rehabilitation Unit of Policlinico Italia Centre, Rome, Italy. Patients were admitted for outpatient rehabilitation between May 2014 and April 2017. All patients were in a stable drug program and had adapted to their current medications for at least 2 weeks.
  All participants could walk independently without walking devices. All patients were taking oral administrations of levodopa (18 patients), dopamine agonists (5 patients), or both (13 patients) and were recorded in on phase. Patients' clinical and anthropometric characteristics.
  Severity of parkinsonism was evaluated using the Unified Parkinson's Disease Rating Scale (UPDRS-II and III) and the Hoehn and Yahr staging system.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
stance duration (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  time interval between two consecutive foot strikes of the same lower limb) expressed as a percentage of the stride duration
step length (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  the distance measured from the heel print of one foot to the heel print of the other foot
Step width (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  Step width variability discriminates gait of healthy young and older adults during treadmill locomotion.
walking speed (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  distance coverde by the body in unit of time
cadence (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  time of steps per unit time
The flexion-extension hips (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
Trunk saggital plane (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
Trunk frotal plane (change) | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale UPDRS Severity of parkinsonism | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  The UPDRS is made up of these sections:
  * Part I: evaluation of mentation, behavior, and mood
  * Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food
  * Part III: clinician-scored monitored motor evaluation
  * Part IV: complications of therapy
Modified Hoehn and Yahr staging | - T0 at baseline before rehabilitative treatment - T1 10- week after rehabilitative treatments
  1. Unilateral involvement only usually with minimal or no functional disability Unilateral involvement only 1.5 - Unilateral and axial involvement
  2. Bilateral or midline involvement without impairment of balance Bilateral involvement without impairment of balance 2.5 - Mild bilateral disease with recovery on pull test
  3. Bilateral disease: mild to moderate disability with impaired postural reflexes; physically independent Mild to moderate bilateral disease; some postural instability; physically independent
  4. Severely disabling disease; still able to walk or stand unassisted Severe disability; still able to walk or stand unassisted
  5. Confinement to bed or wheelchair unless aided Wheelchair bound or bedridden unless aided

CONTACTS AND LOCATIONS:
Overall Officials: Guido Caramanico, MD, Principal Investigator — Università "La Sapienza di Roma"
Locations (1):
- Policlinico Italia Srl, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meunier S, Pol S, Houeto JL, Vidailhet M. Abnormal reciprocal inhibition between antagonist muscles in Parkinson's disease. Brain. 2000 May;123 ( Pt 5):1017-26. doi: 10.1093/brain/123.5.1017. PMID 10775546
- [Background] Pistacchi M, Gioulis M, Sanson F, De Giovannini E, Filippi G, Rossetto F, Zambito Marsala S. Gait analysis and clinical correlations in early Parkinson's disease. Funct Neurol. 2017 Jan/Mar;32(1):28-34. doi: 10.11138/fneur/2017.32.1.028. PMID 28380321
- [Background] Vieregge P, Stolze H, Klein C, Heberlein I. Gait quantitation in Parkinson's disease--locomotor disability and correlation to clinical rating scales. J Neural Transm (Vienna). 1997;104(2-3):237-48. doi: 10.1007/BF01273184. PMID 9203085
- [Background] Pau M, Corona F, Pili R, Casula C, Sors F, Agostini T, Cossu G, Guicciardi M, Murgia M. Effects of Physical Rehabilitation Integrated with Rhythmic Auditory Stimulation on Spatio-Temporal and Kinematic Parameters of Gait in Parkinson's Disease. Front Neurol. 2016 Aug 11;7:126. doi: 10.3389/fneur.2016.00126. eCollection 2016. PMID 27563296
- [Background] Keus SH, Munneke M, Nijkrake MJ, Kwakkel G, Bloem BR. Physical therapy in Parkinson's disease: evolution and future challenges. Mov Disord. 2009 Jan 15;24(1):1-14. doi: 10.1002/mds.22141. PMID 18946880